CLINICAL TRIAL: NCT04570722
Title: Implementing Ipsilateral Peripheral Intravenous Access Procedures for Routine Scanning in Patients With a History of Surgical Axillary Procedures (The iPIVAP Study)
Brief Title: Ipsilateral Peripheral Intravenous Access Procedures (The iPIVAP Study)
Acronym: iPIVAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00106186
Record Dates: First submitted 2020-09-16; First posted 2020-09-30 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Melanoma; Thoracic Cancer; Lymphedema of Upper Arm
MeSH Terms: conditions — Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): Patients with a history of axillary surgical lymph node procedures (SLNP) presenting for routine radiographic scan will complete baseline measures: bilateral volumetric measurements and self-reported symptoms. Patients will undergo SOC contralateral arm intravenous access attempt. After one failed attempt, ipsilateral intravenous access instead of pedal or neck access will be offered per research protocol. Nursing documentation will reflect the failed venipuncture and categorize a reason for the failed attempt.
  Interventions: Other: Ipsilateral peripheral IV insertion

INTERVENTIONS:
Other: Ipsilateral peripheral IV insertion — Patients with successful ipsilateral intravenous access will be provided a patient education sheet describing signs and symptoms that should be reported to the study team. All participants will be contacted by the study team at twelve week intervals for 12 months after their radiology encounter for completion of symptom assessments. If a subject reports new signs or symptoms of lymphedema during follow-up, a clinic appointment for volumetric measurements and thorough evaluation will occur

SUMMARY:
This pilot study will examine facilitators and barriers that impact staff uptake for implementation of practice change involving ipsilateral IV insertion in patients with axillary lymphadenectomy/dissection in a single radiology center.

DETAILED DESCRIPTION:
This prospective single arm study will be conducted within DUH Department of Radiology CT Imaging. The study team will enroll 50 patients with a history of axillary SLNP presenting for routine radiographic scan to undergo ipsilateral IV insertion. Patients will complete baseline bilateral arm volumetric measurements and self-reported symptom assessments. Patients will be followed every 3 months for 1-year duration for development of lymphedema. Patient acceptance or reluctance to ipsilateral IV access will be categorized at time of screening. Staff uptake on practice change will be assessed through medical record documentation for number, location, and factors affecting IV attempts and their perceptions of practice change and acceptance at the end of one year.

All participants will complete baseline measures: bilateral volumetric measurements and self-reported symptoms. Per DUH policy, participants will undergo SOC contralateral arm intravenous access attempt. After one failed attempt, ipsilateral intravenous access instead of pedal or neck access will be offered per research protocol. Nursing documentation will reflect the failed venipuncture and categorize a reason for the failed attempt. At the discretion of the treating radiologist, a participant who has a history of multiple failed IV placement attempts in the contralateral arm may proceed to IV placement in the ipsilateral arm on the first attempt.

Patients with successful ipsilateral intravenous access will be provided a patient education sheet describing signs and symptoms that should be reported to the study team. All participants will be contacted by the study team at twelve week intervals for 12 months after their radiology encounter for completion of symptom assessments. If a subject reports new signs or symptoms of lymphedema during follow-up, a clinic appointment for volumetric measurements and thorough evaluation will occur within 2 weeks; findings will be discussed with their physician. Participants will undergo bilateral volumetric measurements, symptom assessments, and perceptions of the ipsilateral IV access protocol at the end of one year.

ELIGIBILITY:
Inclusion Criteria:

1. History of bilateral or unilateral axillary SLNP (sentinel biopsy, lymphadenectomy or dissection) and a previous or current failed contralateral IV attempt or at the discretion of the treating radiologist, a participant who has a history of multiple failed IV placement attempts in the contralateral arm may proceed to IV placement in the ipsilateral arm on the first attempt
2. Scheduled to undergo routine imaging scan with contrast
3. 18 years of age and older
4. Read, reviewed and signed study-specific consent

Exclusion Criteria:

1. Active swelling, rash, or injury in bilateral upper extremities
2. Subjects with diabetes, sickle cell disease, and/or peripheral vascular insufficiency as vascular inflammatory processes pose a lymphedema risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Identify facilitators and barriers that impact staff uptake for implementation of practice change involving ipsilateral IV insertion in patients with axillary lymphadenectomy/dissection. | Through study completion, an average of 2 years.
  Perceptions of barriers and facilitators by staff will be collected at study end using a qualitative format. Modeled after Melnyk, Fineout-Overholt, and Mays (2008) EBP surveys, open-ended questions will be asked during a focus group to ascertain their perceptions of the impact of the ipsilateral IV access protocol. Staff will be asked what worked well, what barriers did they experience, and what do they recommend for protocol adoption. Constant comparative analysis will be used to categorize themes from their responses

SECONDARY OUTCOMES:
Volumetric measurements | Baseline and at 12 months post ipsilateral IV insertion
  Volumetric measurements will be obtained using a tape measure to assess limb girth circumference at five anatomic points. A difference of 2 centimeters or more in arm circumference at a corresponding point between ipsilateral and contralateral arms is considered a common criterion for a diagnosis of lymphedema.(Armer et al 2003)
Lymphedema symptoms; patient reported outcomes (PRO) | Baseline, every 3 months after intervention for 12 months
  The Lymphedema Breast Cancer Questionnaire (LBCQ) uses 3 items to assess 19 symptoms most commonly associated with lymphedema (Radina et al., 2007). The LBCQ shows an acceptable measure of internal consistency (r=.785) for all 19 items. Test-retest reliability was evaluated using a sample of healthy women without breast cancer or lymphedema (n=35) over a 2-hour test-retest interval. The findings show a high degree of reliability (r =.98).
Self reported lymphedema changes :patient reported outcomes (PRO) | Baseline, every 3 months after intervention for 12 months
  The Lymphedema Scale uses 2 items for self-reported changes in wrist, elbow, and upper arm sizes. Scale sensitivity ranged from 0.86-0.92 in women with circumferential arm differences >2 cm indicating presence of moderate lymphedema (Norman et al., 2001).
Study participation acceptance | Baseline
  Potential participants who decline to enroll at time of phone screening: the study team will ask if they would be willing to share a reason for their reluctance. The reasons will be categorized as qualitative responses at the end of study, for example: "I must ask my oncologist permission, I've been told to never allow a procedure in my affected arm".
  b) For those enrolled: their perceptions regarding the ipsilateral access will be ascertained at the time of quarterly phone follow-up and at the end of study. Qualitative data will be analysed thematically.
  Patient perceptions of acceptance will be assessed in those who opt to or not to participate in thestudy:

CONTACTS AND LOCATIONS:
Overall Officials: Deborah H Allen, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No